CLINICAL TRIAL: NCT01269554
Title: Etiology of Diarrhea in Guinea-Bissau and in Finland
Status: Completed | Type: Observational
Sponsor: Bandim Health Project (Other)
Collaborators: University of Helsinki (Other); Stockholm University (Other)
Responsible Party: Sponsor
Other Study IDs: Diar-GB-Finland 2011
Record Dates: First submitted 2010-11-13; First posted 2011-01-04 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2015-08

CONDITIONS: Diarrhea
Keywords: diarrhea; Guinea-Bissau; Finland; Children; Adults; Intestinal pathogens; Bacteria; Virus; Parasites
MeSH Terms: conditions — Diarrhea; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Faecea samples are collected for analysis of patogens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Children with diarrhea in Bissau
- Children without diarrhea in Bissau
- Children without diarrhea in Finland
- Children with diarrhea in Finland
- Adults without diarrhea in Finland
- Adults with diarrhea in Finland
- Adults without diarrhea in Bissau
- Adults with diarrhea in Bissau

SUMMARY:
Diarrhoea is the leading cause of death in the world with 2.2 million deaths every year. The majority of deaths are among children in developing countries, but the travellers encounter the disease as well. The studies on the aetiology have suffered from serious methodological deficiencies and the results are even controversial. At the same time, the current diagnostic methods are inadequate. The investigators have recently developed novel multiplex RT-PCR methods to cover the majority of diarrhoeal pathogens. The present study is a collaboration between Finland and Sweden/Guinea-Bissau. The aim is to characterize the causative agents of diarrhoea (a) in Finnish volunteers before and after a travel to tropical areas and, (b) in inhabitants of endemic areas in Guinea-Bissau. For these purposes stool samples will be collected from volunteers of different age groups and from healthy volunteers as well as those with diarrhea both in Guinea-Bissau and in Finland. In addition to pathogens, other intestinal microbes and antimicrobial resistance will be investigated

ELIGIBILITY:
Inclusion Criteria:

1. Accepting to participate and willing to deliver 2 stool samples.
2. With diarrhea: the first 10 children and 10 adults presenting each month at the health facility Without diarrhea: In Bissau matched controls drawn from the registration system at Bandim Health Project. In Finland controls selected at the health facilities participating.

Exclusion Criteria:

* Not willing or able to deliver the stool samples

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. children and adults with diarrhea reporting to Bandim Health Centre
  2. age and sex mached children and adults without diarrhea from Bandim
  3. children and adults with a recent travel history and suffering from diarrhea reporting to Postitalo Travel Clinic
  4. children and adults without diarrhea and no recent travel history reporting to Postitalo Travel Clinic
Sampling Method: Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Type of pathogens in stool samples in percentage of included patients | 2 years
  The percentage of included patients with different pathogens will be described.

SECONDARY OUTCOMES:
Type of microbes other than than pathogens in stool samples in percentage of included patients | 2 years
The patern of resistance to antimicrobials in isolated pathogens | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, Ph.d, Principal Investigator — Helsinki University Central Hospital,Dept of Medicine, Division of Infectious Diseases, Aurora Hospital, Building 5, Floor 3, POB 3448, FIN-00029 HUS
Locations (3):
- Finland (2):
  - Postitalo Travel Clinic, Helsinki
  - University of Helsinki, Helsinki
- Bandim Health Centre, Bissau, Guinea-Bissau